CLINICAL TRIAL: NCT01534637
Title: A Feasibility Study to Discern the Tolerability of 5-FU/Gemcitabine Based Chemotherapy Concurrent With Upper Abdominal Radiation and the Utility of Aprepitant/5HT-3 Antagonist (EMEND) for the Prevention of ChemoRadiation-Induced Nausea and Vomiting (CRINV)
Brief Title: Aprepitant in Preventing Nausea and Vomiting in Patients Undergoing Chemotherapy and Radiation Therapy for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00000209; NCI-2009-01258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 02205 (Other: Wake Forest University Health Sciences); NCT00398164 (obsolete NCT alias)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Extrahepatic Bile Duct Cancer; Nausea; Vomiting; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Nausea; Vomiting; Pancreatic Neoplasms | interventions — Aprepitant; Gemcitabine; Capecitabine; Fluorouracil; Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (antiemetic, chemotherapy, and radiation therapy) (Experimental): CHEMORADIOTHERAPY: Patients undergo radiation therapy once daily on days 1-5 for 5.5 weeks. Patients also receive gemcitabine hydrochloride IV over 30 minutes once weekly and either fluorouracil IV continuously or capecitabine PO twice daily on days 1-5.
  PROPHYLACTIC THERAPY: Beginning 1 hour before chemoradiotherapy, patients receive aprepitant PO on days 1-3. Treatment repeats every 7 days for 5.5 weeks in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION CHEMOTHERAPY: Two to four weeks after completion of chemoradiotherapy and prophylactic therapy, patients without disease progression or a declining performance status receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: aprepitant; Drug: gemcitabine hydrochloride; Drug: capecitabine; Drug: fluorouracil; Procedure: radiation therapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: nausea and vomiting therapy; Procedure: management of therapy complications

INTERVENTIONS:
Drug: aprepitant — Given PO
  Other Names: Emend; L-754030; MK-0869; ONO-7436
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Procedure: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Procedure: nausea and vomiting therapy — Receive aprepitant
  Other Names: antiemetic support; management of nausea and vomiting; nausea and vomiting management; therapy, nausea and vomiting; vomiting and nausea management
Procedure: management of therapy complications — Receive aprepitant
  Other Names: complications of therapy, management of

SUMMARY:
This pilot clinical trial is studying how well aprepitant works in preventing nausea and vomiting in patients undergoing chemotherapy and radiation therapy for pancreatic cancer. Antiemetic drugs, such as aprepitant may help lessen or prevent nausea and vomiting in patients receiving chemotherapy and radiation therapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Discern the gastrointestinal toxicities associated with 5-FU (fluorouracil)/Gemcitabine (gemcitabine hydrochloride) chemotherapy when combined with upper abdominal radiation therapy.

II. Determine if the addition of prophylactic Aprepitant/5HT-3/Dexamethasone therapy to standard chemoradiation for patients with pancreatic cancer results in less nausea and vomiting when compared to historical controls.

SECONDARY OBJECTIVES:

I. To determine the impact of prophylactic Aprepitant/5HT-3/Dexamethasone therapy on the impact of emesis on daily living, as measured using the MASCC Antiemesis (MAT) tool.

OUTLINE:

CHEMORADIOTHERAPY: Patients undergo radiation therapy once daily on days 1-5 for 5.5 weeks. Patients also receive gemcitabine hydrochloride intravenously (IV) over 30 minutes once weekly and either fluorouracil IV continuously or capecitabine orally (PO) twice daily on days 1-5.

PROPHYLACTIC THERAPY: Beginning 1 hour before chemoradiotherapy, patients receive aprepitant PO on days 1-3. Treatment repeats every 7 days for 5.5 weeks in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION CHEMOTHERAPY: Two to four weeks after completion of chemoradiotherapy and prophylactic therapy, patients without disease progression or a declining performance status receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of carcinoma arising from the pancreas
* Resected or unresectable pancreatic cancer, potentially resectable, or resectable (neoadjuvant) disease (stage II and III); stage IV patients with symptomatic back pain requiring palliation are also eligible at the discretion of the Principal Investigator (PI); resected patients, i.e. - "Whipple" of biliary ductal cancers are also eligible at the discretion of the PI
* Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Evidence of disease; this can be measurable, evaluable, or nonmeasurable
* Estimated life expectancy of at least 12 weeks
* Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 X 10^9/L
* Platelets >= 100 X 10^9/L
* Hemoglobin >= 9 g/dL
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase (AP) =< 3.0 ULN ( AP =< 5 x ULN is acceptable if liver has tumor involvement)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 ULN (AST and ALT =< 5 x ULN is acceptable if liver has tumor involvement)
* Albumin >= 3.0 g/dL
* Signed informed consent from patient
* Male and female patients with reproductive potential must use an approved contraceptive method (e.g., intrauterine device, birth control pills, or barrier device) during and for 3 months after the study

Exclusion Criteria:

* Active infection (at the discretion of the investigator)
* Neuroendocrine tumor of the pancreas
* Documented brain metastasis; brain imaging in symptomatic patients is required to rule out metastases, but not required in asymptomatic patients
* Pregnancy
* Breast feeding
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Use of any investigational agent within 4 weeks before enrollment into the study
* Significant cardiovascular disease in the form of abnormal electrocardiogram (ECG) coupled with clinical features of recent or recurrent cardiac disease (including myocardial infarction, angina or hypertension)
* Prior treatment with chemotherapy for pancreatic cancer
* Clinically significant effusions (pleural or peritoneal) that cannot be drained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Blackstock, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting patients 08/31/2006 and closed to enrollment 12/03/2009. Patients were recruited from the Comprehensive Cancer Center of Wake Forest Baptist Health.
Period: Overall Study
Arm/Group | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy)
Started | 22
Completed | 13
Not Completed | 9
Not completed — Physician Decision | 3
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Liver Mets before treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Gastrointestinal Toxicities (Grade 3 and 4 Nausea and Vomiting) Associated With Delivering Fluorouracil/Gemcitabine Hydrochloride-based Chemotherapy With Upper Abdominal Radiation
Description: Toxicity will be determined using the revised National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 3.0 for Toxicity and Adverse Event Reporting. Descriptive statistics (means, standard deviations, frequencies, etc.) will be presented for pretreatment patient characteristics. The rate of grade 3 and 4 nausea will be compared to the cut points during interim and final analyses.
Time Frame: Over 10 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy)
Number analyzed (Participants) | 20
participants | 3

2. Secondary Outcome: Impact of Aprepitant/5HT-3 Antagonist Therapy on the Patient Quality of Life as Measured by the Number of Patients Using Anti Nausea Drugs
Time Frame: Week 1
Measure: Number; unit: participants
Arm/Group | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy)
Number analyzed (Participants) | 19
participants | 6

3. Secondary Outcome: Impact of Aprepitant/5HT-3 Antagonist Therapy on the Patient Quality of Life as Measured by the Number of Patients Taking Anti Nausea Drugs
Time Frame: Week 5
Measure: Number; unit: participants
Arm/Group | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy)
Number analyzed (Participants) | 15
participants | 5

ADVERSE EVENTS:
Arm/Group | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 5/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy) (N=21)
Anorexia (Gastrointestinal disorders) | 1 (1) — Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); IV fluids, tube feedings or TPN indicated
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Pain: Abdomen (Nervous system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Antiemetic, Chemotherapy, and Radiation Therapy) (N=21)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (4) — 4 non serious (grade 1 or 2) occurrances
Platelets (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
Nausea (Blood and lymphatic system disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) — 2 non serious (grade 1-2) occurances
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 4 (4) — 4 non serious (grade 1-2) occurances
Albumin, serum-low (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2/2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes